CLINICAL TRIAL: NCT03659227
Title: Adverse Cutaneous Drug Reactions Collection of Clinical Data and Biological Samples
Brief Title: Drug Reactions Sampling (COLLECTIONTOXIDERMIES)
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K180201J
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Stevens-Johnson Syndrome; Lyell Syndrome; Drug Reactions; AGEP; DRESS; Bullous Dermatosis Caused by Drug Treatment (Disorder); Maculopapular Exanthem; Erythema Multiforme
Keywords: Drug reactions; severe cutaneous adverse reactions (SCARs; Stevens-Johnson syndrome; Lyell Syndrome; (generalized bullous) fixed drug reaction; AGEP; DRESS; drug induced IgA bullous dermatosis; maculopapular exanthema; erythema multiforme; sampling; collection
MeSH Terms: conditions — Stevens-Johnson Syndrome; Drug-Related Side Effects and Adverse Reactions; Drug Eruptions; Erythema Multiforme; Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * one skin punch biopsy
  * blood (serum, cells, DNA and RNA studies);
  * blister fluid aspiration;
  * oral and nose mucous membrane and skin eSWABs ;
  * stool samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intro: Dermatology department of Henri Mondor Hospital (Creteil, France), is a reference center for toxic bullous diseases and severe cutaneous drug reactions (Stevens-Johnson syndrome (SJS), Lyell syndrome (toxic epidermal necrolysis (TEN)), generalized bullous fixed drug reactions, AGEP, DRESS, drug induced immunoglobulin A (IgA) bullous dermatosis, and erythema multiforme). In order to conduct clinical and biological research studies in drug reactions, it is necessary for the investigator's department to implement a collection of clinical data and biological samples.

Hypothesis/Objective: To collect clinical data and cutaneous and biological samples for immunological, biological and genetic studies to improve knowledge about pathophysiology of drug reactions.

Method: The following samples will be performed in addition to the routine practice samples: one skin punch biopsy (6mm); 43 mL of blood; blister fluid aspiration; oral and nose mucous membrane and skin eSWABs, stool samples.

These samples will be stored in a dedicated biological sampling department ("Platform of biological resources").

Conclusion: The implementation of this collection should allow us to conduct pathophysiological studies about drug reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 y-old
* Severe cutaneous drug reaction (AGEP, DRESS, SJS/TEN, generalized bullous fixed drug eruption), drug-induced IgA bullous dermatosis, maculopapular exanthema, erythema multiforme
* Signed consent
* Social security affiliation

Exclusion Criteria:

* Patients law protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe cutaneous adverse reactions (DRESS, AGEP, SJS/TEN, generalized bullous fixed drug eruption), drug-induced IgA linear dermatosis, maculo-papular exanthema, erythema multiforme.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-09-25 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
Implementation of a clinical data and biological samples collection for cutaneous adverse reactions | Day 0
  Implementation of a clinical data and biological samples collection for cutaneous adverse reactions

SECONDARY OUTCOMES:
To conduct clinical and biological (immunological, histological, microbiological and genetic) studies in cutaneous adverse reactions. | Day 0
  To conduct clinical and biological (immunological, histological, microbiological and genetic) studies in cutaneous adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Oro, MD, Principal Investigator — APHP
Locations (1):
- Henri Mondor, Créteil, France